CLINICAL TRIAL: NCT04851470
Title: Periodontal Assessment of a Bariatric Care Population, Clinical, Genetic and Microbiological Characteristics. A Cross-sectional Study.
Brief Title: Periodontal Assessment of a Bariatric Care Population
Acronym: Bariatric
Status: Recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS ID 108243
Record Dates: First submitted 2021-03-08; First posted 2021-04-20 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Bariatric Surgery Candidate; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples of Saliva, Dental bacterial Plaque and Venous Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our primary aim is to investigate the prevalence and severity of Periodonotal Disease (PD) in a population of obese patients.

Our secondary objectives are to:

Investigate inflammatory biomarkers that have been associated with PD in the saliva of obese patients.

Investigate the association of FTO gene (Obesity) polymorphisms with the prevalence of PD in this population.

Investigate and describe the subgingival microbial flora in obese patients with PD from subgingival dental plaque samples as well as the salivary samples.

DETAILED DESCRIPTION:
Overall design and plan of the study This is a cross-sectional association study. The study population will be recruited among individuals attending the UCLH Centre for Weight Loss, Metabolic & Endocrine Surgery (UCLH bariatric clinic) and have given written informed consent to the study.

Experimental Design All individuals who consent to this study will receive as part of their routine care a medical examination, where a series of parameters are recorded (including age, gender, smoking status, Bio-impedance for full body composition, ethnicity, and body mass index). These data will be copied for this study. A blood sample will also be collected for genetic analysis unless the patients have DNA already collected and it has been verified that the results are available. In that case no venepuncture will be needed.

All subjects will receive a basic periodontal examination (BPE). For individuals with signs of destructive periodontitis (BPE scores 3-4) full mouth plaque and gingival bleeding scores will also be calculated. In addition to that also a comprehensive full mouth periodontal probing depths assessment will be performed.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all of the following inclusion criteria to be enrolled in the study:

1. Subject must be over 18 years of age.
2. Subject must have a BMI of higher or equal to 30 kg/ m2
3. Subject must have voluntarily given written informed consent.

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria are not to be enrolled in the study:

1. Subject is currently involved in other research involving the use of antibiotics or novel or unknown medications.
2. Self-reported pregnancy.
3. Subject is on chronic treatment (i.e., two weeks or more) with specific medications known to affect periodontal status (phenytoin or cyclosporine) within one month of baseline visit.
4. Subject knowingly has HIV or Viral Hepatitis.
5. Patients are completely edentulous.
6. Subject with uncontrolled systemic illnesses.
7. Subject is not capable to give informed consent.
8. Subjects on chronic antibiotic therapy (ie two weeks or more in the previous month).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a cross-sectional association study. The study population will be recruited among individuals attending the UCLH Centre for Weight Loss, Metabolic & Endocrine Surgery (UCLH bariatric clinic) and have given written informed consent to the study.
Sampling Method: Probability Sample
Enrollment: 394 (Estimated)
Dates: Start 2014-01-31 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Periodontal Disease in an Obese Population | Cross-sectional study, single visit study so only one time point. Up to two hours from consent to obtain the BPE examination and full mouth periodontal examination.
  Basic Periodontal Examination (BPE) scores and full mouth periodontal examination. BPE scores are given per sextant of the mouth and they can take values of 0 to 4 and or asterisk.

SECONDARY OUTCOMES:
Investigation of inflammatory biomarkers that have been previously been associated with Periodontal Disease in the saliva of obese patients. | Cross-sectional study, single visit study so only one time point at the collection of the salivary sample. Up to two hours from consent to obtain the sample.
  Salivary samples aliquots will be analysed with Elisa or Multiplex assay for a series of human inflammatory markers of interest. The results of the quantitative analysis will be combined with the clinical findings to investigate for correlation with the periodontal disease status of the patients.
Correlation of FTO gene (Obesity) polymorphisms with the prevalence of PD in obese population | Cross-sectional study, single visit study so only one time point at the collection of the blood sample.Up to two hours from consent to obtain the sample.
  DNA will be extracted from venepunctured blood and will be genotyped for the FTO polymorphism at position rs9939609. The presence of the rare allele will be analysed with the clinical findings to investigate for correlation with the periodontal disease status of the patients.
Correlation of subgingival microbial flora in obese patients with and without periodontitis. | Cross-sectional study, single visit study so only one time point at the collection of the sample. Up to two hours from consent to obtain the sample.
  Salivary samples aliquots and subgingival bacterial samples will be used for extraction and genotyping of bacterial DNA using high throughput sequencing. Bioinformatics will be used to correlate between periodontal disease status and bacterial microbiome.

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Donos, Prof., Principal Investigator — Professor of Periodontology and Implantology
Locations (4):
- United Kingdom (4):
  - Barts Health NHS Trust Dental Hospital, London
  - Centre for Oral Clinical Research (COCR), London
  - St Bartholomew's Hospital, Barts Health NHS Trust, London
  - Luton and Dunstable University Hospital, Luton